CLINICAL TRIAL: NCT03378817
Title: Hypothermic Oxygenated Machine Perfusion of Extended Criteria Kidney Allografts From Brain Death Donors - a Prospective Cohort Study
Brief Title: Hypothermic Oxygenated Machine Perfusion of Extended Criteria Kidney Allografts From Brain Death Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Responsible Party: Principal Investigator, Georg Lurje, M.D., Attending Transplant Surgeon, University Hospital, Aachen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 184-17
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Reperfusion Injury; Hypothermic Oxygenated Machine Perfusion
Keywords: Extended criteria donor; Donation after brain death; HOPE; Kidney transplantation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: Pilot study, case matched (1:2)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional cold storage (Active Comparator): Conventional static cold storage (CCS) on temperature 0-4 °C from organ procurement (historical case matched group)
  Interventions: Other: Conventional cold storage
- Hypothermic oxygenated perfusion (HOPE) (Experimental): HOPE for 1 hour via the renal artery in a recirculating and pressure controlled system, Belzer (UW) machine perfusion solution, perfusate temperature 0-4 °C, perfusate oxygenation pO2 of 60-80 kPa Other Name: Hypothermic machine perfusion (HMP)
  Interventions: Procedure: HOPE

INTERVENTIONS:
Procedure: HOPE — HOPE for 1 hour via the renal artery in a recirculating and pressure controlled system, Belzer (UW) machine perfusion solution, perfusate temperature 0-4 °C, perfusate oxygenation pO2 of 60-80 kPa Other Name: Hypothermic machine perfusion (HMP)
  Arms: Hypothermic oxygenated perfusion (HOPE)
Other: Conventional cold storage — No intervention
  Arms: Conventional cold storage

SUMMARY:
Kidney transplantation (KT) has emerged as the mainstay of treatment for end-stage kidney disease. In an effort to address the widening gap between demand and supply of donor organs, there has been an increase in the numbers of "marginal" or functionally impaired renal allografts that had to be accepted for KT over the decades. The use of extended criteria donor (ECD) allografts is associated with a higher incidence of primary graft non-function (PNF) and/or delayed graft function (DGF). Hypothermic oxygenated machine perfusion (HOPE) has been successfully tested in pre-clinical experiments and in a few clinical series of donation after cardiac death (DCD) in liver transplantation. The present trial is an investigator-initiated pilot study on the effects of HOPE on ECD-allografts in donation after brain death (DBD) KT. Fifteen kidney allografts will be submitted to 2 hours of HOPE before implantation and are going to be compared to a case matched group transplanted after conventional cold storage (CCS).

DETAILED DESCRIPTION:
The present trial is an investigator-initiated pilot study on the effects of HOPE on ECD-allografts in DBD KT. Fifteen kidney allografts with defined inclusion/exclusion criteria will be submitted to 2 hours of HOPE via the renal artery before implantation and are going to be compared to a case matched group of 30 patients (1:2 matching) transplanted after CCS. Besides the clinical evaluation of HOPE-"reconditioned" allograft function, a targeted biomarker analysis is planned using tissue, serum, and urine samples as the translational and basic research aspect of the present study.

ELIGIBILITY:
Inclusion Criteria:

Dialysis-requiring Patients, suffering from end stage kidney disease, listed for KT and receiving ECD organs at the Department of Surgery and Transplantation, University Hospital RWTH Aachen, Aachen, Germany. Informed consent is obtained from all subjects participating in the trial by a qualified member of the study team.

ECD is defined as followed: deceased donors > 60 years and older, and those aged between 50-59 years with at least two of the following conditions: cerebrovascular cause of death, serum Creatinine greater than 1.5 mg/dL (132.6 µmol/L), history of arterial hypertension

Exclusion Criteria:

1. Recipients of living donor kidney transplants
2. Previous kidney transplantation
3. Participation in other kidney related trials
4. The subject received an investigational drug within 30 days prior to inclusion
5. The subject is unwilling or unable to follow the procedures outlined in the protocol
6. The subject is mentally or legally incapacitated
7. Non-German or non-English speakers
8. Family members of the investigators or employees of the participating department
9. The subject is mentally or legally incapacitated
10. The subject suffers from uncontrolled bacterial or viral infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
DGF | 7 days post-transplant
  DGF (defined as the need for dialysis in the first 7-days post-transplantation)

SECONDARY OUTCOMES:
CRR2, CRR5 | 5 days post-transplant
  Creatinine reduction ratio day 2 (CRR2= creatinine day 1-creatinine day 2/creatinine day 1) and CRR5 (CRR5=pre-transplant creatinine-creatinine day 5/pre-transplant creatinine)
postoperative complications | Subjects will be followed 6 months postoperatively
  Clavien-Dindo complication score
Cumulative postoperative complications | Subjects will be followed 6 months postoperatively
  Comprehensive complication index (CCI)
Duration of intensive care stay | Subjects will be followed 6 months postoperatively
  Duration of ICU stay
Duration of hospital stay | Subjects will be followed 6 months postoperatively
  Duration of hospitalisation
Graft survival | Subjects will be followed 6 months postoperatively
  Six months graft survival
Renal function | Subjects will be followed 6 months postoperatively
  Renal function (serum creatinine and estimated glomerular filtration rate (eGFR))
Perfusion Parameter | During HOPE
  Flow and thus renal resistance

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lurje, M.D., Principal Investigator — RWTH Aachen University
Locations (1):
- Department of Surgery and Transplantation, University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meister FA, Czigany Z, Rietzler K, Miller H, Reichelt S, Liu WJ, Boecker J, Moeller MJ, Tolba RH, Hamesch K, Strnad P, Boor P, Stoppe C, Neumann UP, Lurje G. Decrease of renal resistance during hypothermic oxygenated machine perfusion is associated with early allograft function in extended criteria donation kidney transplantation. Sci Rep. 2020 Oct 20;10(1):17726. doi: 10.1038/s41598-020-74839-7. PMID 33082420
- [Derived] Meister FA, Czigany Z, Bednarsch J, Bocker J, Amygdalos I, Morales Santana DA, Rietzler K, Moeller M, Tolba R, Boor P, Rohlfs W, Neumann UP, Lurje G. Hypothermic Oxygenated Machine Perfusion of Extended Criteria Kidney Allografts from Brain Dead Donors: Protocol for a Prospective Pilot Study. JMIR Res Protoc. 2019 Oct 14;8(10):e14622. doi: 10.2196/14622. PMID 31613224